CLINICAL TRIAL: NCT02581852
Title: Workability in Patients With Seropositive Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Franz Josef Hospital (Other)
Collaborators: Landsteiner Institut (Other)
Responsible Party: Principal Investigator, Carolin Berner, Prof. Dr. Ludwig Erlacher, Kaiser Franz Josef Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Workability in RA
Record Dates: First submitted 2015-07-10; First posted 2015-10-21 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Seropositive Rheumatoid Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm assessment (Other): Cross sectional assessment of workability, functional disability, frailty, muscle strength, quality of sleep and sexual functioning of rheumatoid arthritis patients with different disease activity levels.
  Interventions: Other: Cross sectional assessment

INTERVENTIONS:
Other: Cross sectional assessment — Assessment of workability, functional disability, frailty, muscle strength, quality of sleep and sexual functioning

SUMMARY:
This study compares workability in subjects with seropositive rheumatoid arthritis (RA) in the working age with high and low disease activity. Further interest is to clarify the influence of frailty, functional ability and muscle strength on workability and to determine the effect of disease activity on selected physiological needs (sleep quality, sexual functioning). Methods include a physical examination, questionnaires and physical tests.

DETAILED DESCRIPTION:
Chronic diseases like RA are negatively associated with workability and RA has been shown to be an economic burden for society and patients. RA patients seem also to be more prone to frailty which is characterized by slowed walking speed, low physical activity, and low grip strength. Also poor sleep has been shown to negatively influence work ability and the majority of patients with RA experience insomnia, general fatigue and mental fatigue. RA has also been shown affect sexual functioning.

This monocentric cross sectional study will be conducted at a Viennese rheumatological outpatient clinic and day hospital on about 100 seropositive RA patients. The primary objective of this study is to compare workability in subjects with seropositive RA in the working age with high and low disease activity. Secondary interest is to clarify the influence of frailty, functional ability and muscle strength on workability and to determine the effect of disease activity on selected physiological needs (sleep quality, sexual functioning). Disease activity will be assessed during the patient's routine visit at the clinic via the clinical disease activity index (CDAI). Workability will be determined by the Work Ability Index questionnaire. The influencing determinants frailty and functional disability will be also assessed via questionnaires and/or with physical examinations (Survey of Health, Ageing and Retirement in Europe Frailty instrument, Short Physical Performance Battery, Health Assessment Questionnaire-Disability Index). For muscle strength assessment hand grip and maximum quadriceps strength will be measured . Contributing physiologic needs quality sleep and sexual functioning will be additionally determined vial self reported questionnaire (Medical Outcome Study -Sleep Scale, Index for sexual functioning).

In order to compare patients with low and high disease activity regarding metric data (like sleep quality or sexual functioning) unpaired Students t-tests (given normal distributed data and homogeneous variances), Welch corrected unpaired Student t-tests (in case of normal distributed data but heterogenous variances) or Mann-Whitney-U tests (in case of skewed data) will be used. Kolmogorov-Smirnov and Levene tests will be used to test for normal distribution and homogenous variances.To assess the impact of frailty, functional ability, muscle strength on workability (high versus low) binary logistic regression will be applied. In general the alpha level is set to 5%.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive rheumatoid arthritis according to EULAR Criteria
* Age ≥18 and ≤65 years

Exclusion Criteria:

* Cannot understand questionnaires in the languages provided (German , English, Turkish, Serb o-Croatian)
* Cannot understand instructions for physical tests/assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Workability | Day 1
  Self-reported work ability will be measured by the work ability index (WAI). The WAI is a questionnaire consisting of seven subscales: current work ability compared with the lifetime best; work ability in relation to the demands of the job; number of current diseases diagnosed by a physician; estimated work impairment due to disease; sick leave during the past 12 month; own prognosis of work ability 2 years from now; and mental resources. The cumulative index of WAI ranges from 7 to 49 points. It is then divided into 4 categories: poor (7-27 points), moderate (28-36 points), good (37-43 points) and excellent work ability (44-49 points).

SECONDARY OUTCOMES:
Functional Disability | Day 1
  Extend of the patients´ self-reported functional disability will be assessed by the Health Assessment Questionnaire Disability Index (HAQ -DI). There are 20 questions in eight categories of functioning - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Self-reported difficulties to perform these activities are scored on a scale from 0 to 3, representing normal (no difficulty) (0), some difficulty (1), much difficulty (2), and unable to do (3). For any component question, highest score determines the score for that respective domain. The overall disability index is a value between 0 ( no functional disability) and 3 (severe functional disability) representing the average score across the domains.
Frailty | Day 1
  Frailty will be assessed with the SHARE Frailty Instrument (SHARE- FI).The assessment comprises 5 variables: grip strength measurement and 4 questions related to weakness, exhaustion, slowness and the activity level. Using the 5 variables DFactor scores (DFS) will be calculated using the gender specific SHARE-FI formula. For each subject the frailty score will be computed and subjects will then be categorized as non-frail, pre-frail, or frail.
Lower-extremity function | Day 1
  Lower-extremity function will be measured with the short physical performance battery (SPPB). The SPPB is a group of measures including gait speed, chair stand and balance tests. Each test a five-level categorical score will be assessed, with 0 representing inability to complete the test and 4 representing the highest level of performance. The summary score ranges from 0 (worst performance) to 12 (best performance).
Musculus quadriceps femoris strength | Day1
  Quadriceps muscle strength will be measured with an isokinetic dynamometer.Strength will be assessed 3 times for both legs with a 2 minute break between the measurements. Per software analysis maximum peak value of every leg will be determined on the basis of power vs. time curve. Mean value of both legs will be used in the statistical analysis.
Hand grip strength | Day1
  Maximum grip strength will be measured with a portable hydraulic hand dynamometer. Three maximum voluntary grip strength contractions will be taken for each hand. Measurements will be done in alternating order with a 2 minutes break between each measurement. The mean value of each hand will be taken for analysis.
Quality of sleep | Day1
  The patients´ quality of sleep will be assessed with the MOS Sleep Scale (MOS -SS) questionnaire.The MOS-SS is a 12-item self -report questionnaire referring to a retrospective assessment over the past 4 weeks. The MOS measures 6 sleep dimensions: Initiation (time to fall asleep in minutes), quantity (hours of sleep each night), maintenance, respiratory problems, perceived adequacy and somnolence. The last 4 items will be assessed via a 6-item scale ranging from "all the time" to "none of the time". The questionnaire yields 2 sleep problem indexes and 6 scores.
Sexual functioning | Day1
  Sexual functioning will be measured via self-assessment questionnaire individually designed for this study.The questionnaire consists of two sections addressing sexual disability (difficulties in performing sexual intercourse) represented by question 1 and sexual drive ( reflected in sexual desire and satisfaction) represented by question 2-5. Scoring ranges from 1-10 and anchor points are set according to the question. Overall sexual functioning score ranges from 5 points (poor sexual functioning) to max 50 points.

OTHER OUTCOMES:
IL-6 | Day1
  IL-6 levels will be measured in the blood. Standard venous blood sampling.
TNF-alpha | Day1
  TNF-alpha levels will be measured in the blood. Standard venous blood sampling.
CRP | Day 1
  CRP-alpha levels will be measured in the blood. Standard venous blood sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dorner, Assoc Prof, MD, MPH, Study Chair — Institute of Social Medicine and Centre of Public Health; Ludwig Erlacher, Prof. MD, Principal Investigator — Kaiser Franz Josefs Hospital

REFERENCES:
- [Derived] Berner C, Erlacher L, Quittan M, Fenzl KH, Dorner TE. Workability and Muscle Strength in Patients With Seropositive Rheumatoid Arthritis: Survey Study Protocol. JMIR Res Protoc. 2017 Mar 2;6(3):e36. doi: 10.2196/resprot.6449. PMID 28254736